CLINICAL TRIAL: NCT04563780
Title: The Prognostic Value of Post Thyroidectomy 99mTCpertechnetate Thyroid Scan in Patient With Differentiated Thyroid Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Khaled Mahmoud, resident doctor, Assiut University
Other Study IDs: 99mTC thyroid scan in DTC
Record Dates: First submitted 2020-09-21; First posted 2020-09-24 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Differentiated Thyroid Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: 99mTC pertechnetate thyroid scan — Thyroid scintigraphy was performed just before RIT. 20 min after intravenous injection 99mTc-pertechnetate, anterior images of the neck were acquired using a scintillation camera equipped with low-energy high resolution collimator. Energy discrimination was provided with a 20% window that was centered on the 140 keV peak of 99mTc .

SUMMARY:
The aim of this study is to evaluate the prognostic value of postoperative99mTc-pertechnetate scanning in patients with DTC.

DETAILED DESCRIPTION:
The incidence of thyroid cancer in several affluent countries has markedly increased (1). Although mortality from thyroid cancer has remained relatively low and stable or has steadily declined in these and other countries (2).

Therefore, it is still important to identify markers for prognosis prediction and decision-making before radioactive iodine therapy (RIT). Various factors have been reported to be associated with the clinical outcome of RIT. These include preablative stimulated thyroglobulin (ps- Tg), tumor size, extrathyroidal invasiveness, cervical lymph node metastasis and TSH [3,4].

99mTc pertechnetate is a radiopharmaceutical used for thyroid scintigraphy. The photon energy of 140kev is ideally suited for use with gamma camera. It has short half life of about 6-hoursand no particulate emissions. 99mTc-pertechnetate scintigraphy is a simple, economic and RIT non-interfering technique to evaluate the volume of residual thyroid tissue(RTT). The 99m Tc-pertechnetate uptake of the thyroid bed can be used as a marker of RTT. Although negative uptake doesn't indicate the absence of RTT, it could suggest a small volume. On the other hand, positive uptake can be considered as a large volume of RTT. Several studies have reported that patients with negative 99mTc-pertechnetate uptake have a much higher chance of successful ablation[5, 6].

We hypothesized that negative 99mTc-pertechnetate scintigraphy is a significant predictor for excellent response (ER) to RIT in American Thyroid Association 2015(ATA) low- and intermediate risk DTC patient according to .

ELIGIBILITY:
Inclusion Criteria:

* • This study will include pathologically proved DTC patients in low and intermediate risk according to ATA who presented to nuclear medicine unit during the period from 2015 until the end of the study.

Exclusion Criteria:

* • High risk patient according to ATA

  * Pregnancy

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all patient underwent total thyroidectomy in low and intermediate risk will done thyroid scan
Sampling Method: Non-Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The prognostic value of post thyroidectomy 99mTCpertechnetate thyroid scan in patient with differentiated thyroid cancer | baseline
  The prognostic value of post thyroidectomy 99mTCpertechnetate thyroid scan in patient with differentiated thyroid cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Aya Khaled Mahmoud, Asyut, Egypt

REFERENCES:
- [Background] Dal Maso L, Panato C, Franceschi S, Serraino D, Buzzoni C, Busco S, Ferretti S, Torrisi A, Falcini F, Zorzi M, Cirilli C, Mazzucco W, Magoni M, Collarile P, Pannozzo F, Caiazzo AL, Russo AG, Gili A, Caldarella A, Zanetti R, Michiara M, Mangone L, Filiberti RA, Fusco M, Gasparini F, Tagliabue G, Cesaraccio R, Tumino R, Gatti L, Tisano F, Piffer S, Sini GM, Mazzoleni G, Rosso S, Fanetti AC, Vaccarella S; for AIRTUM working group. The impact of overdiagnosis on thyroid cancer epidemic in Italy,1998-2012. Eur J Cancer. 2018 May;94:6-15. doi: 10.1016/j.ejca.2018.01.083. Epub 2018 Mar 20. PMID 29502036
- [Background] Li M, Brito JP, Vaccarella S. Long-Term Declines of Thyroid Cancer Mortality: An International Age-Period-Cohort Analysis. Thyroid. 2020 Jun;30(6):838-846. doi: 10.1089/thy.2019.0684. Epub 2020 Mar 2. PMID 31964280
- [Background] Liu N, Meng Z, Jia Q, Tan J, Zhang G, Zheng W, Wang R, Li X, Hu T, Upadhyaya A, Zhou P, Wang S. Multiple-factor analysis of the first radioactive iodine therapy in post-operative patients with differentiated thyroid cancer for achieving a disease-free status. Sci Rep. 2016 Oct 10;6:34915. doi: 10.1038/srep34915. PMID 27721492
- [Background] Jung JS, Lee SM, Kim SJ, Choi J, Han SW. Prediction of the success of thyroid remnant ablation using preablative 99mTc pertechnetate scintigraphy and postablative dual 131I scintigraphy. Nucl Med Commun. 2015 Jan;36(1):38-44. doi: 10.1097/MNM.0000000000000219. PMID 25299469
- [Background] Tsai CJ, Cheng CY, Shen DH, Kuo SJ, Wang LY, Lee CH, Wang JJ, Chang MC, Huang WS. Tc-99m imaging in thyroidectomized differentiated thyroid cancer patients immediately before I-131 treatment. Nucl Med Commun. 2016 Feb;37(2):182-7. doi: 10.1097/MNM.0000000000000426. PMID 26626550
- [Background] Furuya-Kanamori L, Bell KJL, Clark J, Glasziou P, Doi SAR. Prevalence of Differentiated Thyroid Cancer in Autopsy Studies Over Six Decades: A Meta-Analysis. J Clin Oncol. 2016 Oct 20;34(30):3672-3679. doi: 10.1200/JCO.2016.67.7419. PMID 27601555